CLINICAL TRIAL: NCT04308551
Title: Effect of Indobufen and Aspirin on Platelet Aggregation and Long Term Prognosis in Patients With Stable Coronary Heart Disease. A Prospective, Randomized and Controlled，Single Blind, Single-center, Opening Study
Brief Title: Effect of Indobufen and Aspirin on Platelet Aggregation and Long Term Prognosis in Patients With Coronary Heart Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: shortage of funds
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HenanICE202001
Record Dates: First submitted 2020-03-06; First posted 2020-03-16 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Stable Coronary Heart Disease
MeSH Terms: interventions — indobufen; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The treatment in this study was open. Optical density turbidimetric platelet aggregation (LTA) and thromboelastography (TEG) were used to detect the platelet aggregation rate induced by AA and ADP, and the metabolites were measured by ELISA. All were done by the laboratory personnel, and they were unaware of the setting of treatment medication (blind method).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indobufen (Experimental): 200 mg Indobufen, bid po, 90 days
  Interventions: Drug: Indobufen
- Aspirin (Active Comparator): 100 mg Aspirin, qd po, 90 days
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Indobufen — Indobufen Tablets
  Arms: Indobufen
Drug: Aspirin — Aspirin Tablets
  Arms: Aspirin

SUMMARY:
This study evaluates the effect of Indobufen and Aspirin on platelet aggregation and long term prognosis in patients with stable coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years < age ≤ 85 years;
2. Patients with confirmed stable coronary heart disease (must meet at least one of the following conditions);

   2.1 a stenosis confirmed by Coronary angiography or dual-source CT, but the stenosis of the Left Main Artery (LMA) diameter is less than 50%, the stenosis of the left anterior descending branch（LAD）is less than 70%, and the stenosis of the two or three coronary arteries diameter is less than 70%, patient has no corresponding evidence of ischemia;

   2.2 Patients after percutaneous coronary intervention (PCI): Dual antiplatelet therapy (DAPT) time is greater than 9 months, without cardiovascular events and ischemic symptoms; and currently receiving aspirin 100 mg/d with clopidogrel 75 mg/d or ticagrelor 90mg (bid) dual antiplatelet therapy.

   2.3 Patients after coronary artery bypass graft (CABG): Dual antiplatelet therapy (DAPT) time is greater than 9 months, without cardiovascular events and ischemic symptoms; and currently receiving aspirin 100 mg/d with clopidogrel 75 mg/d or ticagrelor 90mg (bid) dual antiplatelet therapy.
3. Willing to sign the informed consent.

Exclusion Criteria:

1. Acute coronary syndrome (ACS) occurred within 3 months before screening;
2. Percutaneous coronary intervention or CABG surgery within 9 months before screening;
3. Any other conditions (such as atrial fibrillation, pulmonary embolism, lower extremity venous thrombosis, artificial heart valve, etc.) who need oral or intravenous anticoagulation treatment;
4. In the past 3 months, the Arachidonic acid-induced platelet aggregation rate≥ 50%; inhibition rate ≤ 20% in the aspirin combined with clopidogrel treated patients;
5. Congestive heart failure or left ventricular ejection fraction <35%;
6. A positive history of Chronic Obstructive Pulmonary Disease (COPD);
7. bleeding tendency or severe lung disease;
8. Active pathological bleeding;
9. History of intracranial hemorrhage (less than 3 months);
10. Allergic to indobufen / aspirin (or any of its ingredients);
11. Severe liver injury (transaminases exceeding the upper limit of 2 times and above);
12. Pregnancy, lactation and those who have a birth plan;
13. Hematological diseases, platelet count <100000 / mm3 or hemoglobin <10g / dL;
14. Have a history of drug or alcohol abuse in the past 2 years;
15. Use of non-steroidal anti-inflammatory drugs (within 3 months);
16. Creatinine clearance <30ml/min;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Arachidonic acid and Adenosine diphosphate-induced platelet aggregation rates 7 days after taking the Indobufen or Aspirin | 7 days
  Patients with stable coronary heart disease were treated with Indobufen or Aspirin for 90 days. Subsequently, the investigators used the Light transmission aggregation(LTA) and Thrombelastography (TEG) methods to detect the Arachidonic acid and Adenosine diphosphate-induced platelet aggregation rates on the 7 days.
Arachidonic acid and Adenosine diphosphate-induced platelet aggregation rates 30 days after taking the Indobufen or Aspirin | 30 days
  Patients with stable coronary heart disease were treated with Indobufen or Aspirin for 90 days. Subsequently, the investigators used the Light transmission aggregation(LTA) and Thrombelastography (TEG) methods to detect the Arachidonic acid and Adenosine diphosphate-induced platelet aggregation rates on the 30 days.
Arachidonic acid and Adenosine diphosphate-induced platelet aggregation rates 90 days after taking the Indobufen or Aspirin | 90 days
  Patients with stable coronary heart disease were treated with Indobufen or Aspirin for 90 days. Subsequently, the investigators used the Light transmission aggregation(LTA) and Thrombelastography (TEG) methods to detect the Arachidonic acid and Adenosine diphosphate-induced platelet aggregation rates on the 90 days.
Concentration of Thromboxane B2 (TXB2) at baseline | baseline
  The fasting blood was collected after the subjects signed informed consent；And the concentration of TXB2 was detected by enzyme-linked immuno sorbent assay (ELISA)
Concentration of Thromboxane B2 (TXB2) 7 days after taking the Indobufen or Aspirin | 7 days
  The fasting blood was collected 7 days after taking the Indobufen or Aspirin；And the concentration of TXB2 was detected by enzyme-linked immuno sorbent assay (ELISA)
Concentration of Thromboxane B2 (TXB2) 30 days after taking the Indobufen or Aspirin | 30 days
  The fasting blood was collected 30 days after taking the Indobufen or Aspirin；And the concentration of TXB2 was detected by enzyme-linked immuno sorbent assay (ELISA)
Concentration of Thromboxane B2 (TXB2) 90 days after taking the Indobufen or Aspirin | 90 days
  The fasting blood was collected 90 days after taking the Indobufen or Aspirin；And the concentration of TXB2 was detected by enzyme-linked immuno sorbent assay (ELISA)

SECONDARY OUTCOMES:
Incidence of Bleeding | baseline, 7, 30 and 90 days
  During the study period, we used dual occult blood and questionnaire format to assess whether the subject experienced bleeding (the extent and location of the bleeding) and the degree of bleeding related to indobufen or aspirin (Certainly, likely, possible, suspicious, impossible)
Incidence of Adverse Gastrointestinal reaction | 7, 30 and 90 days
  During the study period, we used dual occult blood and questionnaire format to assess whether the subject experienced adverse gastrointestinal reaction, such as nausea, vomiting, upper abdominal discomfort or pain, gastric mucosal damage, gastric ulcers and bleeding, etc
Blood concentration | 7, 30 and 90 days
  The fasting blood was collected on the day of 7 days, 30 days, and 90 days；And the blood concentration of aspirin or indobufen or clopidogrel or ticagrelor was detected.
Cyclooxygenase-1 gene phenotype | baseline
  The fasting blood was collected and saved on the day of enrollment, and then the gene phenotype of cyclooxygenase-1 would be detected, and their relationship with platelet aggregation also would be analyzed.
Major adverse cardiovascular events | 7, 30 and 90 days
  Number of angina pectoris symptoms, non ST-segment elevation myocardial infarction (NSTEMI), ST-segment elevation myocardial infarction (STEMI), stroke, cardiovascular death, cerebrovascular death, all-cause death

CONTACTS AND LOCATIONS:
Overall Officials: chuanyu gao, MD, Principal Investigator — central china fuwai hospital

IPD SHARING:
Plan to Share IPD: No